CLINICAL TRIAL: NCT01678209
Title: Imaging Stimulant and Non Stimulant Treatments for ADHD: A Network Based Approach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Newcorn, Director Division of Child and Adolescent Psychiatry, Associate Professor Psychiatry and Pediatrics, Medical Director Center for Excellence for ADHD and Related Disorders, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 11-0161; 5R01MH095766-02 (NIH)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; ADHD
Keywords: Attention Deficit Hyperactivity Disorder; Stimulant; Non-stimulant; Drug; Methylphenidate; Atomoxetine; Strattera; Concerta; MACRO; Medication; Treatment; Youth; Adolescent; Functional Magnetic Resonance Imaging; Brain scan; Imaging; Response inhibition; Inattentive; Hyperactive; Combined; Medication Treatment; Brain Imaging
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm | interventions — Atomoxetine Hydrochloride; Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fMRI scans (Active Comparator): Healthy Control Group: will receive initial evaluation, and 2 fMRI (functional magnetic resonance imaging) scans each 6-8 weeks apart
  Interventions: Other: fMRI scans
- Atomoxetine arm (Experimental): These subjects will receive initial evaluation and baseline fMRI scan, flexible dose titration with atomoxetine for 6-8 weeks, and fMRI postscan, with optional post study stabilization visits.
  Interventions: Other: fMRI scans; Drug: Atomoxetine arm
- Methylphenidate arm (Experimental): Subjects will receive initial evaluation, baseline fMRI scan, flexible dose titration with methylphenidate (Concerta) for 6-8 weeks, and fMRI scan post treatment.
  Interventions: Other: fMRI scans; Drug: Methylphenidate arm

INTERVENTIONS:
Other: fMRI scans — 2 fMRI scans 6-8 weeks apart
Drug: Atomoxetine arm — Flexible dose titration with atomoxetine prescribed at weekly visits for 6-8 weeks
  Other Names: Strattera; ATX
  Arms: Atomoxetine arm
Drug: Methylphenidate arm — Flexible dose titration with methylphenidate for 6-8 weeks, with optional post study stabilization visits.
  Other Names: Concerta; MPH
  Arms: Methylphenidate arm

SUMMARY:
The growing number of medications used to treat attention-deficit/hyperactivity disorder (ADHD) raises important questions about whether different medications have similar or different therapeutic mechanisms of action. We have recently shown that the stimulant methylphenidate (MPH) and the non-stimulant atomoxetine (ATX) produce clinical improvement via a common mechanism in motor cortex, and distinct actions in frontostriatal and midline cingulate-precuneus regions. These exciting findings offer a window into the common and unique neurophysiological mechanisms of response to stimulant and non-stimulant treatments. However, the interpretation and clinical utility of these results would be greatly enhanced by in-depth investigation of the impact of the two treatments on relevant neural networks, and analyses which evaluate whether improvement is achieved via normalization or other adaptive changes in brain function.

DETAILED DESCRIPTION:
The specific aims of this project are to use functional magnetic resonance imaging (fMRI) to determine the significance of activation changes over treatment related to clinical improvement, and the impact of treatment on neural connectivity within and between the anti-correlated frontostriatal 'task-positive' circuit and cingulate-precuneus 'task-negative' network. Our central hypotheses are that clinical improvement is associated with: (i) normalization of reduced connectivity of regions within the 'task-positive' network, with resultant increased inhibition of motor cortex, and (ii) normalization of low task-related connectivity in regions within the task-negative network for MPH and the 'task-positive' network for ATX.

This research proposes to test a model which posits a neurophysiological basis of mechanisms of response to stimulant and non-stimulant medications, and fits with our long term objectives of being able to match treatments to individual patients. Testing this model requires large samples of youth scanned using fMRI before and after treatment, and matched healthy controls also scanned twice. We will use an innovative network-based approach to study the effects of treatment, building on results from our current fMRI treatment study, and incorporating new theoretical approaches to understanding ADHD and its treatment.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria for subjects with ADHD and healthy controls are:

* aged 7-17 years;
* Wechsler Intelligence Scale for Children (WISC) scores ≥ 75;
* informed consent and assent to study participation.

Specific inclusion criteria for youth with ADHD are:

* diagnosis of ADHD, any subtype, determined by Kiddie Schedule for Affective Disorders and Schizophrenia for School-Aged Children-Present and Lifetime Versions (K-SADS-PL);
* ADHD Rating Scale-IV-Parent Version: Investigator Administered (ADHD-RSIV) total score ≥ 1.5 SD above age and gender means for subtype
* Clinical Global Impressions-ADHD-Severity (CGI-S) score > 4;
* ADHD must be the primary diagnosis and focus of treatment, and the treatments offered in the study must not be contraindicated for the comorbid disorder.

Exclusion Criteria:

General exclusion criteria are:

* history of head injury with loss of consciousness or any CNS disease that is likely to affect brain function;
* diagnosis of autism or pervasive developmental, psychotic, major mood, and Tourette's disorder;
* alcohol or drug abuse in the past 3 months or a positive urinary toxic screen on initial evaluation;
* use of psychotropic medication within 2 weeks of the study (8 weeks for fluoxetine);
* pre-existing medical or psychological condition which precludes being in the scanner (e.g., claustrophobia, morbid obesity);
* metal in the body that precludes scanning (e.g., braces, metal plate);
* positive urine pregnancy test.

Specific exclusion criteria for the treatment trial include:

* previous unsuccessful trial of MPH or ATX that was adequately dosed (≥ 1 mg/kg for MPH or 1.0 mg/kg for ATX) and of adequate duration (≥ 4 weeks);
* abnormal findings on physical exam, or vital signs
* pulse and blood pressure > 95% of age and gender mean;
* inability to swallow capsules;
* weight is < 20 kg or > 85 kg.

Specific exclusion criteria for control youth include:

* no past history or current diagnosis of any psychiatric disorder, determined by the K-SADS-PL interview;
* ADHD-RS-IV and CBCL scores for each symptom domain ≤ 1 SD of age and gender means.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2012-10; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Newcorn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Kurt Schulz, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: 8/10/2012 - 4/30/17; Roll Over Year: 5/1/17 - 4/30/18; Youth with ADHD and Healthy Controls recruited from the community and clinics at Mount Sinai.
Groups:
- Control Group fMRI Scans Only: Healthy Control Group: will receive initial evaluation, and 2 fMRI (functional magnetic resonance imaging) scans each 6-8 weeks apart
Period: Overall Study
Arm/Group | Control Group fMRI Scans Only | Atomoxetine Arm | Methylphenidate Arm
Started | 47 | 40 | 40
Completed | 30 | 22 | 22
Not Completed | 17 | 18 | 18
Not completed — could not scan twice | 1 | 1 | 1
Not completed — scheduling conflicts | 0 | 0 | 1
Not completed — screen fail | 16 | 17 | 16

BASELINE CHARACTERISTICS:
Population: Only participants with usable data were included in the data results
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group fMRI Scans Only | Atomoxetine Arm | Methylphenidate Arm | Total
Number analyzed (Participants) | 47 | 22 | 22 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 13 (2.8) | 10 (3.02) | 12 (2.86) | 11 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 6 | 27
  Male | 32 | 16 | 16 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 11 | 40
  Not Hispanic or Latino | 32 | 8 | 11 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 3 | 6 | 25
  White | 12 | 4 | 3 | 19
  More than one race | 16 | 14 | 12 | 42
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correct Inhibition in Participants Assessed With the Go-No go Task
Description: Comparison of Go-Nogo at 6 weeks from baseline. Performance on a go-nogo task inside the scanner (fMRI). In the go/no-go task, participants respond to certain stimuli ("go" stimuli) and make no response for others ("no-go" stimuli).
Time Frame: Baseline and at 6 weeks
Population: All participants in control group including the one subject who could not be scanned twice included in data analysis for the 6 weeks visit. Thirty-one (N=31) controls were scanned twice for this project, but the second scan data for 1 subject was excluded from the analysis for motion. Thus, 31 control subjects were included in the analyses of
Measure: Mean (Standard Deviation); unit: percent correct inhibition
Arm/Group | Control Group fMRI Scans Only | Atomoxetine Arm | Methylphenidate Arm
Number analyzed (Participants) | 47 | 40 | 40
percent correct inhibition
  Baseline | 79.08 (15.07) | 79.43 (17.27) | 77.98 (15.10)
  6 weeks: number analyzed (Participants) | 31 | 22 | 22
  6 weeks | 78.24 (16.57) | 80.72 (14.22) | 81.81 (14.14)

2. Secondary Outcome: Adult Attention Deficit Hyperactivity Disorder Investigator Symptom Rating Scale (ADHD-RS)
Description: ADHD-RS is an 18-item list of core ADHD symptoms, each item are scored on a 4-point scale from 0-3, with total 0-54, with higher score indicating more symptoms.
Time Frame: 8 weeks
Population: All participants in control group including the one subject who could not be scanned twice included in data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group fMRI Scans Only | Atomoxetine Arm | Methylphenidate Arm
Number analyzed (Participants) | 31 | 22 | 22
score on a scale | 1 (2) | 15 (11) | 18 (12)

3. Secondary Outcome: Clinical Global Impressions-Severity (CGI-S)
Description: a clinician rated measure of symptom severity. CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: up to 6 weeks
Population: All participants in control group including the one subject who could not be scanned twice included in data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group fMRI Scans Only | Atomoxetine Arm | Methylphenidate Arm
Number analyzed (Participants) | 31 | 22 | 22
score on a scale | 1 (0) | 3.2 (1.6) | 3.4 (1.2)

4. Secondary Outcome: Response Time in Attention Networks Test (ANT)
Description: A neuropsychological assessment of attention compared at 6 weeks from baseline by looking at response time. The ANT is a task designed to test three attentional networks in children and adults: alerting, orienting, and executive control. The response time were summed.
Time Frame: baseline and at 6 weeks
Population: All participants in control group including the one subject who could not be scanned twice included in data analysis for the 6 weeks visit.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Control Group fMRI Scans Only | Atomoxetine Arm | Methylphenidate Arm
Number analyzed (Participants) | 47 | 40 | 40
milliseconds
  Baseline | 817.50 (171.06) | 856.60 (179.34) | 885.68 (170.76)
  6 weeks: number analyzed (Participants) | 31 | 22 | 22
  6 weeks | 756.87 (153.83) | 826.14 (139.08) | 783.09 (125.21)

5. Secondary Outcome: Continuous Performance Test (CPT)
Description: A neuropsychological assessment of attention compared at 6 weeks from baseline. CPT is a task-oriented computerized assessment of attention-related problems.This score indicates the number of times the client responded but no target was presented. A fast reaction time and high commission error rate points to difficulties with impulsivity. A slow reaction time with high commission and omission errors, indicates inattention in general. Scores are compared with the normative scores for the age, group and gender of the person being tested and represented as a commissioned T-score. The T-score indicates the degree to which performance in CPT task is higher or lower than the performance of a healthy individual matched in age. A T-score of 50 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of more attention-related problems.
Time Frame: baseline and at 6 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: commissioned t-score
Arm/Group | Control Group fMRI Scans Only | Atomoxetine Arm | Methylphenidate Arm
Number analyzed (Participants) | 47 | 40 | 40
commissioned t-score
  Baseline | 46.65 (11.29) | 55.26 (5.62) | 52.94 (9.19)
  6 weeks: number analyzed (Participants) | 31 | 22 | 22
  6 weeks | 44.64 (9.70) | 50.70 (8.66) | 48.46 (10.43)

6. Secondary Outcome: Digit Span
Description: A cognitive/neuropsychological measure of auditory/verbal working memory compared at 6 weeks from baseline. Digit Span. Memory span is the longest list of items that a person can repeat back in correct order immediately after presentation on 50% of all trials. Items may include words, numbers, or letters. The task is known as digit span when numbers are used. Memory span is a common measure of short-term memory. A digit-span task is used to measure working memory's number storage capacity.The item score is the sum of the scores on the two trials for that item (range=0-2). The total raw score for backwards digit span is the sum of the item scores; maximum backwards digit span total raw score is 0-16 points. Higher score indicates better health outcomes.
Time Frame: baseline and at 6 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group fMRI Scans Only | Atomoxetine Arm | Methylphenidate Arm
Number analyzed (Participants) | 47 | 40 | 40
score on a scale
  Baseline | 13.30 (18.76) | 9.25 (2.06) | 7.5 (1.29)
  6 weeks: number analyzed (Participants) | 31 | 22 | 22
  6 weeks | 9.39 (1.58) | 9.75 (0.95) | 8.5 (1.29)

7. Secondary Outcome: Finger Windows
Description: A neuropsychological measure of motor skill and visual-spatial working memory compared at 6 weeks from baseline. The Finger Windows subtest is a measure of nonverbal, rote sequential recall. scaled scores ranging from 1 to 19, with higher score indicating better attention or concentration.
Time Frame: baseline and at 6 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group fMRI Scans Only | Atomoxetine Arm | Methylphenidate Arm
Number analyzed (Participants) | 47 | 40 | 40
score on a scale
  Baseline | 17.04 (3.69) | 14.50 (2.64) | 16.50 (5.19)
  6 weeks: number analyzed (Participants) | 31 | 22 | 22
  6 weeks | 17.65 (5.33) | 16.25 (6.65) | 16.25 (6.39)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | fMRI Scans | Atomoxetine Arm | Methylphenidate Arm
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 3/47 | 6/22 | 4/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | fMRI Scans (N=47) | Atomoxetine Arm (N=22) | Methylphenidate Arm (N=22)
Decreased appetite (Gastrointestinal disorders) | 0 | 2 | 4
Stomachache (Gastrointestinal disorders) | 0 | 3 | 1
Headache (General disorders) | 0 | 2 | 1
Moody/irritable (Psychiatric disorders) | 1 | 3 | 3
Common cold/allergies (General disorders) | 1 | 1 | 4
Anxious (Psychiatric disorders) | 0 | 0 | 1
Sleep problems (General disorders) | 2 | 4 | 1
Lightheaded/dizzy (General disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Increased blood pressure (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Dr. Newcorn has FCOI reporting obligations as stipulated by the Mount Sinai FCOI committee

DOCUMENTS (2):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT01678209/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT01678209/SAP_001.pdf